CLINICAL TRIAL: NCT04822298
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 160 in Subjects With Non-Small Cell Lung Cancer
Brief Title: Study of AMG 160 in Subjects With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen made a business decision to discontinue AMG 160 20180273
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180273
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer; NSCLC
Keywords: AMG 160; Phase 1b
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Exploration (Experimental): The dose exploration part of the study will estimate the MTD and/or the RP2D.
  Interventions: Drug: AMG 160
- Part 2: Dose Expansion - Cohort 1 Non-squamous NSCLC (Experimental): Participants with non-squamous non-small cell lung cancer (NSCLC) will be administered the RP2D identified from the dose exploration part of the study.
  Interventions: Drug: AMG 160
- Part 2: Dose Expansion - Cohort 2 Squamous NSCLC (Experimental): Participants with squamous NSCLC will be administered the RP2D identified from the dose exploration part of the study.
  Interventions: Drug: AMG 160

INTERVENTIONS:
Drug: AMG 160 — AMG 160 administered as an intravenous (IV) infusion

SUMMARY:
This study aims to evaluate the safety and tolerability of AMG 160 and to evaluate the maximum tolerated dose (MTD) or the recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Histologically or cytologically confirmed stage 4 or recurrent non-squamous NSCLC (Part 1); histologically or cytologically. confirmed stage 4 or recurrent NSCLC (Part 2 only, squamous cell histology/cytology allowed in Part 2).
* Without a driver mutation: disease progression following at least one line of prior chemotherapy and at least 1 prior anti-programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PDL1) therapy.
* With a driver mutation must experience disease progression on at least 1 targeted therapeutic agent to be eligible.
* Detectable prostate-specific membrane antigen (PSMA) expression by PSMA positron emission tomography (PET)/computed tomography (CT) imaging.
* Measurable disease by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0- 2.

Exclusion Criteria:

* Radiographic evidence of intratumor cavitation, major blood vessel invasion or encasement by cancer.
* Untreated or symptomatic brain metastases and leptomeningeal disease.
* History of hemoptysis within 3 months prior to first dose.
* History or evidence of gastrointestinal inflammatory bowel disease (ulcerative colitis or Crohn disease).
* Myocardial infarction, unstable angina, cardiac arrhythmias requiring medication, and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months prior to start of dosing.
* Vasculitis or grade 3/4 gastrointestinal bleeding within 3 months prior to first dose; vascular disease (eg, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months of first dose.
* Gastrointestinal (GI) perforation and/or fistulae within 6 months prior to start of dosing.
* Interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with treatment.
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
* Chronic systemic corticosteroid therapy or any other immunosuppressive therapies unless stopped 7 days prior to first dose.
* Any biological therapy or immunotherapy within 3 weeks of start of first dose.
* Major surgery within 4 weeks of first dose.
* Infection requiring IV antimicrobials for management within 7 days of dosing.
* Known human immunodeficiency virus (HIV) infection, hepatitis C infection.
* Active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Chris OBrien Lifehouse, Camperdown, New South Wales, Australia
- Austria (2):
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in Australia and Austria between 31 August 2021 and 26 January 2022.
Pre-assignment Details: The study was terminated early due to sponsor decision after 3 participants were enrolled into Cohort 1 of Part 1 (dose exploration); no participants were screened or enrolled for additional Part 1 or Part 2 (dose expansion) cohorts.
Groups:
- Part 1: AMG 160 Cohort 1: AMG 160 was administered as a short-term intravenous (IV) infusion every 2 weeks after the target dose was reached. Treatment lasted until disease progression, up to a planned maximum of 3 years from the first dose of AMG 160.
Period: Overall Study
Arm/Group | Part 1: AMG 160 Cohort 1
Started | 3
Completed | 0
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set: defined as all participants that were enrolled and receive at least 1 dose of AMG 160.
Groups:
- Part 1: AMG 160 Cohort 1: AMG 160 was administered as a short-term IV infusion every 2 weeks after the target dose was reached. Treatment lasted until disease progression, up to a planned maximum of 3 years from the first dose of AMG 160.
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience One or More Dose-limiting Toxicities (DLT)
Description: DLT were defined as any adverse event (AE) with an onset within first 28 days following first dose of AMG 160 meeting pre-specified criteria unless clearly attributable to causes other than AMG 160 treatment.
Time Frame: Day 1 to Day 28
Population: DLT analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160 with an evaluable DLT endpoint. The DLT endpoint is evaluable if either: 1) the participant experienced a DLT, or 2) the participant did not experience a DLT after receiving all planned doses within the 28-day DLT window.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Participants | 1

2. Primary Outcome: Number of Participants Who Experience One or More Treatment-emergent AE (TEAE)
Description: An AE is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. A TEAE is any AE that occurred on or after first dose of study treatment up to 30 days after the last dose or End of Study date or start of new anti-cancer therapy, whichever is earlier. A treatment-related TEAE is any TEAE that, per investigator review, has a reasonable possibility of being caused by the study treatment.
  Any abnormal vital signs measurement or clinical laboratory test result, including those that worsened from Baseline, that were considered clinically significant in the medical and scientific judgement of the investigator were reported as an AE.
Time Frame: Median (min, max) time from first dose to 30 days after the last dose, end of study or start of new anti-cancer therapy; whichever is earlier, was 66 (52, 100) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least 1 dose of AMG 160.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Participants
  Any TEAEs | 3
  Any treatment-related TEAEs | 3

3. Secondary Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR per modified RECIST v1.1 was defined as the percentage of participants who achieved a best overall response (BOR) of either complete response (CR) or partial response (PR) based on investigator assessment.
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm.
  * PR: Decrease of 30% or greater in tumor burden compared with baseline.
  CR/PR must have been confirmed at least 4 weeks later.
  Exact 95% confidence interval (CI) was calculated using the Clopper-Pearson method.
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: RECIST v1.1 evaluable analysis set: defined as all participants that are enrolled, receive at least 1 dose of AMG 160 and had measurable baseline disease per RECIST 1.1 per protocol and had the opportunity to be followed for at least 9 weeks starting from study Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Percentage of Participants | 0.0 [0.00 to 70.76]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of study Day 1 until death due to any cause. OS time (months) = (date of death - study Day 1 + 1) x 12/365.25.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and percentiles were using Greenwood's formula to estimate the standard error of the landmark estimates using the method by Kalbfleisch and Prentice (1980).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Months | 3.29 [3.09 to NA] — Upper limit of the 95% CI was not reached.

5. Secondary Outcome: Radiographic Progression Free Survival (PFS) Per Modified RECIST v1.1
Description: Radiographic PFS per modified RECIST v1.1 was defined as the interval from study Day 1 to the earlier of a radiographic progressive disease (PD) or death from any cause, based on investigator assessment; otherwise, radiographic PFS was censored at the last evaluable tumor assessment date.
  - PD: Increase of 20% or greater in tumor burden compared with nadir and at least 5 mm absolute increase, or unequivocal progression of non-target lesions, or the presence of new lesions.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and quartiles were estimated using the method by Brookmeyer and Crowley (1982).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Months | 3.29 [1.51 to NA] — Upper limit of the 95% CI was not reached.

6. Secondary Outcome: Clinical PFS Per Modified RECIST v1.1
Description: Clinical PFS per modified RECIST v1.1 was defined as the interval from study Day 1 to the earlier of a clinical PD or death from any cause, based on investigator assessment; otherwise, clinical PFS was censored at the last evaluable tumor assessment date.
  - PD: Increase of 20% or greater in tumor burden compared with nadir and at least 5 mm absolute increase, or unequivocal progression of non-target lesions, or the presence of new lesions.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and quartiles were estimated using the method by Brookmeyer and Crowley (1982).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Months | 3.09 [3.09 to NA] — Upper limit of the 95% CI was not reached.

7. Secondary Outcome: Time to Response Per Modified RECIST v1.1
Description: Time to response per modified RECIST v1.1 was defined as the interval from study Day 1 to the either CR or PR based on investigator assessment.
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm.
  * PR: Decrease of 30% or greater in tumor burden compared with baseline.
  CR/PR must have been confirmed at least 4 weeks later.
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160. Analyzed in participants with an objective response.
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Progression Per Modified RECIST v1.1
Description: Time to progression per modified RECIST v1.1 was defined as the interval from study Day 1 to PD, based on investigator assessment. Time to progression was censored at the last evaluable post-baseline tumor assessment prior to subsequent anti-cancer therapy; otherwise at study Day 1.
  - PD: Increase of 20% or greater in tumor burden compared with nadir and at least 5 mm absolute increase, or unequivocal progression of non-target lesions, or the presence of new lesions.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and quartiles were estimated using the method by Brookmeyer and Crowley (1982).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Months | 3.29 [1.51 to NA] — Upper limit of the 95% CI was not reached.

9. Secondary Outcome: Time to Clinical Progression
Description: Time to clinical progression was defined as the interval from study Day 1 to PD. Time to clinical progression was censored at the last evaluable post-baseline tumor assessment prior to subsequent anti-cancer therapy; otherwise at study Day 1.
  - PD: Increase of 20% or greater in tumor burden compared with nadir and at least 5 mm absolute increase, or unequivocal progression of non-target lesions, or the presence of new lesions.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and quartiles were estimated using the method by Brookmeyer and Crowley (1982).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 3
Months | NA [3.09 to NA] — Median and upper limit of the 95% CI were not reached.

10. Secondary Outcome: Duration of Response (DOR) Per Modified RECIST v1.1
Description: DOR was defined as the time from the date of an initial objective response per modified RECIST v1.1 to the earlier of soft-tissue progression or death based on investigator assessment.
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm.
  * PR: Decrease of 30% or greater in tumor burden compared with baseline.
  CR/PR must have been confirmed at least 4 weeks later. Participants who had not ended their response at the time of analysis had DOR censored at their last evaluable tumor assessment by CT/MRI scan.
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: RECIST v1.1 evaluable analysis set: defined as all participants that are enrolled, receive at least 1 dose of AMG 160 and had measurable baseline disease per RECIST 1.1 per protocol and had the opportunity to be followed for at least 9 weeks starting from study Day 1. Analyzed in participants with an objective response.
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 0

11. Secondary Outcome: Time to Subsequent Therapy
Description: Time to subsequent therapy was defined as the time from study Day 1 to the time a participant started/received the subsequent cancer therapy/subsequent therapy; otherwise time to subsequent therapy was censored at the last known date of any of the study assessment prior to initiating the subsequent cancer therapy/subsequent therapy.
  Subsequent therapy was defined any anti-cancer therapies intended to treat NSCLC, or any other anti-cancer therapies started after ending study treatment and prior to End of Study.
  Medians and quartiles were estimated using the Kaplan-Meier method. 95% CIs for medians and quartiles were estimated using the method by Brookmeyer and Crowley (1982).
Time Frame: Median (min, max) time from first dose to end of study was 100 (94, 122) days
Population: Safety analysis set: defined as all participants that were enrolled and receive at least one dose of AMG 160. Analyzed in participants who received subsequent therapy.
Arm/Group | Part 1: AMG 160 Cohort 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: median (min, max) time from enrollment to end of study was 106 (97, 126) days. AEs: median (min, max) time from first dose to 30 days after the last dose, end of study or start of new anti-cancer therapy; whichever is earlier, was 66 (52, 100) days.
Description: Serious AEs and other AEs are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study.
Arm/Group | Part 1: AMG 160 Cohort 1
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: AMG 160 Cohort 1 (N=3)
Uveitis (Eye disorders) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: AMG 160 Cohort 1 (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Eyelid oedema (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 3
Conjunctivitis (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT04822298/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT04822298/SAP_001.pdf